CLINICAL TRIAL: NCT04983316
Title: Operative or Nonoperative Management of Tibial Plateau Fractures? Application of Machine Learning Algorithms to Assist in Treatment Decision
Brief Title: TPF Machine Learning Algorithms
Status: Terminated | Type: Observational
Why Stopped: Not enough capacity for recruitment
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Harm Hoekstra, prof. dr., Prof. dr. Harm Hoekstra, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S64352
Record Dates: First submitted 2021-07-16; First posted 2021-07-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Tibial Plateau Fracture
MeSH Terms: conditions — Tibial Plateau Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To adopt a machine learning technique to decide whether operative or non-operative treatment will result in the best patient-outcome.

DETAILED DESCRIPTION:
The overall goal is to adopt a machine learning technique to decide whether operative or non-operative treatment will result in the best patient-outcome.

The primary objectives are to identify the most suitable machine learning algorithm to predict the best treatment for future patients. Whether conservative or operative treatment will lead to the best patient outcome, will be decided on the predicted KOOS score. Several input factors, such as treatment (conservative or operative), number of fracture fragments, location of the fracture, soft tissue involvement,…for each patient will be used as training data for the algorithm. Some of these input data will be derived from CT-scans. Therefore, the CT scans will be segmented in Mimics, for which UZ Leuven recently purchased licenses. The output variable of the training data will be the KOOS score of each patient. Based on the input and output variable, the algorithm will determine a relation between these. For future patients of which the input variable are known, the output variable (=KOOS score) will be predicted both in case of operative and conservative treatment. We hypothesize that the prediction will be improved by adding more input data over time.

To secondary objective is to identify clinical and radiological factors that help predicting the best treatment for future patients.

As an outlook, the machine learning technique could be implemented in the future in clinical practice and utilized as a patient-specific planning tool for tibial plateau fracture management by aiding the surgeon to select the best treatment for a given case. The collected data in this registry will be used to validate the machine learning model. Patients will not yet be treated based on the results of the developed model, the trauma surgeon is responsible to decide which treatment option is best for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Proximal tibia plateau fracture
* Patient is able to attend follow-up visits

Exclusion Criteria:

* Age < 18 years
* Bilateral fractures
* Neurologic disorders (ie paraplegia, CVA, dementia etc.)
* Not understanding Dutch or English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of UZ Leuven
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Machine learning algorithm | 1 year
  To identify the most suitable machine learning algorithm that predicts the best treatment for future patients. The prediction will be improved over time by additional input.

SECONDARY OUTCOMES:
Clinical factors | 1 year
  To identify clinical factors that help predicting the best treatment for future patients
Radiological factors | 1 year
  To identify radiological factors that help predicting the best treatment for future patients

CONTACTS AND LOCATIONS:
Overall Officials: Harm Hoekstra, Prof. MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium